CLINICAL TRIAL: NCT03754608
Title: Validating Imaging Biomarkers of Small Vessel Disease in Diabetic Individuals Using Advanced MRI Techniques.
Status: Completed | Type: Observational
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Other Study IDs: 2000023733
Record Dates: First submitted 2018-10-16; First posted 2018-11-27 (Actual); Last update posted 2021-04-19 (Actual); Status verified 2021-04

CONDITIONS: Small Vessel Disease of Diabetes Mellitus
MeSH Terms: conditions — Diabetic Angiopathies | interventions — Diffusion Tensor Imaging

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood tests are performed on all participants at three time points. When permission exists we are banking CSF and blood products.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Diabetics/No cognitive impairment: These are individuals with diabetes who do not have vascular cognitive impairment as determined by VASCOG criteria.
  Interventions: Diagnostic Test: MRI including cf-MRI, DTI, ASL and CVR.
- Diabetics with vascular cognitive impairment: These are individuals with diabetes who have vascular cognitive impairment as determined by VASCOG criteria.
  Interventions: Diagnostic Test: MRI including cf-MRI, DTI, ASL and CVR.

INTERVENTIONS:
Diagnostic Test: MRI including cf-MRI, DTI, ASL and CVR. — A paradigm developed at Yale University called Cognitive Predictive Modelling which takes connectivity data and reduces it to two smaller network which predict higher and lower performance in a particular task for which these networks have been optimized. This will be supplemented by MRI vascular measures.
  Other Names: Neuropsychological testing (Cantab), basic laboratory blood tests, small number of CSF

SUMMARY:
To develop a set of biomarkers for imaging of small vessel disease in diabetic individuals using advanced MRI techniques. With this the investigators want to document progression of disease both radiologically and clinically.

DETAILED DESCRIPTION:
The investigators will use a paradigm developed at Yale University called Cognitive Predictive Modelling (CPM) which takes connectivity data and reduces it to two smaller network which predict higher and lower performance in a particular task for which these networks have been optimized. Vascular measures will complement this measure.

ELIGIBILITY:
Inclusion Criteria:

A - Vascular cognitive impairment:

1. Presence of diabetes
2. The International Society of Vascular Behavioral and Cognitive Disorders (VASCOG) criteria for vascular cognitive impairment
3. Age between 55 and 90 (inclusive)
4. Score on the Montreal Cognitive Assessment (MOCA) 15 to 23
5. Presence of a responsible caregiver who will accompany mild cognitive impaired (MCI) subjects to all procedures.
6. Evidence of vascular disease
7. The patient should have a capacity to consent.
8. English speakers

B- Cognitively normal elderly Subjects:

1. Presence of diabetes
2. Absence of National Institute on Aging (NIA) - Alzheimer's Association core clinical criteria for probable Alzheimer's Disease (AD) and VASCOG criteria for vascular cognitive impairment.
3. Objective memory scores within normal range for age (do not meet MCI Subjects criterion 2)
4. Age between 55 and 90 (inclusive)
5. English speakers

Exclusion Criteria:

1. Any significant neurologic disease (other than vascular cognitive disease and stroke), such as Parkinson's disease, brain tumor, seizure disorder, multiple sclerosis, or history of significant head trauma followed by persistent neurologic deficits.
2. Any significant systemic disease including hepatic failure, heart failure, renal failure, Chronic obstructive pulmonary disease (COPD), active infection and autoimmune disease.
3. Any significant systemic illness or unstable medical condition, including: uncontrolled or insulin-dependent diabetes mellitus, uncorrected hypothyroidism or hyperthyroidism, or systemic cancer.
4. Investigational agents are prohibited 4 weeks prior to entry and for the duration of the study. Previous treatment with an investigational small molecule with anti-amyloid properties or passive immunization against amyloid within 1 year of study entry. Previous treatment with an active immunization against amyloid.
5. History of schizophrenia or other major psychiatric disorder (DSM IV criteria).
6. History of alcohol or substance abuse or dependence (DSM IV criteria) within the past 2 years.
7. Pregnancy, as determined by screening pregnancy tests for pre-menopausal females
8. Impairment of visual or auditory acuity sufficient to interfere with study procedures.
9. Education level < 6 years.
10. Presence of pacemakers, aneurysm clips, artificial heart valves, ear implants, metal fragments or foreign objects in the eyes, skin or body. The presence of claustrophobia, precluding MRI.
11. Drink more than 5 alcoholic drinks per week or any heavy drinking days in the last 30 days
12. Women who are pregnant or nursing, or fail to use one of the following methods of birth control unless she or partner is surgically sterile or she is postmenopausal (hormone contraceptives [oral, implant, injection, patch, or ring], contraceptive sponge, double barrier [diaphragm or condom plus spermicide], or intrauterine device (IUD)

Ages: 55 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Our study population are those with type 2 diabetes in mid-life and old age, who may or may not have cognitive deficits, whose cognitive deficits (when present) cannot be better explained by other factors. We exclude those who are unable to have MRI or cognitive testing due to a variety of reasons.
Sampling Method: Non-Probability Sample
Enrollment: 63 (Actual)
Dates: Start 2018-11-07 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2020-08-31 (Actual)

PRIMARY OUTCOMES:
Diagnostic Odds ratio for the MRI vascular cognitive impairment biomarker. | 2 years
  This will be calculated from the sensitivity and specificity as compared to clinical diagnosis.

SECONDARY OUTCOMES:
Correlation between the biomarker and cognition | 18 months.
  Assess whether the biomarker can predict the severity of the cognitive performance.

CONTACTS AND LOCATIONS:
Overall Officials: Arash Salardini, MD, Principal Investigator — Yale University
Locations (1):
- Yale University School of Medicine, New Haven, Connecticut, United States